CLINICAL TRIAL: NCT06350604
Title: Project WHADE: A Partner-Based Physical Activity Program for Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-2023-355
Record Dates: First submitted 2024-03-15; First posted 2024-04-05 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2024-11

CONDITIONS: Hypertension; Type 2 Diabetes; Metabolic Syndrome; Smoking; High Cholesterol; PreDiabetes; Prehypertension
Keywords: Social support; Physical activity
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Metabolic Syndrome; Smoking; Hypercholesterolemia; Prediabetic State; Prehypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Project WHADE: A Partner-Based Physical Activity Program for Women (Experimental): Behavioral and cognitive skills to promote physical activity behavior
  Interventions: Behavioral: Project WHADE: A Partner-Based Physical Activity Program for Women

INTERVENTIONS:
Behavioral: Project WHADE: A Partner-Based Physical Activity Program for Women — Combination of behavioral, cognitive, social, and acceptance-based skills training to increase physical activity

SUMMARY:
This study is designed to test the feasibility and acceptability of a new method for supporting physical activity among women ages 40-65 who have risk factors for cardiovascular disease. Each participant receives a trained physical activity coach and a physical activity partner; the partner is another woman in the program. Partners communicate with each other between weekly coaching sessions to provide support for physical activity behavior change.

DETAILED DESCRIPTION:
The purpose of this study is to test the feasibility and acceptability of a new method for supporting physical activity in women ages 40-65 who have risk markers for cardiovascular disease. The primary goal is to understand perceptions of support and communication patterns between partner dyads of women in midlife (ages 40-65). The creation of these partner dyads is a promising method for promoting social support and physical activity for this population. Understanding how partners communicate with one another throughout this intervention study will give insight into how women in this population maximize benefits from partnership through communication and shared experiences (e.g., age, gender, cardiovascular disease risk, interest in being more physically active).

ELIGIBILITY:
Inclusion Criteria:

* One or more of the following health conditions: smoking (current or quit in the last 3 months), or a physician diagnosis of prediabetes or type 2 diabetes, prehypertension or hypertension (high blood pressure), hypercholesterolemia or hyperlipidemia(high cholesterol), or metabolic syndrome
* Engaging in less in less than 6500 steps per day or less than 90 minutes of structured exercise per week
* Access to personal mobile device
* Fluent in English

Exclusion Criteria:

* Pregnant or intend to become pregnant in the next 9 weeks,
* Medical or psychiatric situation that hinders the ability to perform physical activity
* None one of the following cardiovascular risk behaviors or conditions: smoking, diagnosed prediabetes/type 2 diabetes, prehypertension/hypertension, high cholesterol, or metabolic syndrome
* Not fluent in English,
* No access to a personal mobile device

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identification as a woman
Enrollment: 62 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Frequency of partner communication | up to 8 weeks
  How frequently each partner dyad communicates with each other between coaching sessions, assessed via self-report in end of day survey (measure created for this study)
Satisfaction with partner communication | up to 8 weeks
  How satisfied each participant is with their partner communication between coaching sessions, assessed via self-report in end of day survey (measure created for this study)

SECONDARY OUTCOMES:
Physical activity behavior - steps | up to 8 weeks
  Steps per day, assessed with an activity monitor (pedometer with accelerometer)
Physical activity behavior - active minutes | up to 8 weeks
  Minutes of moderate to vigorous activity per day, assessed with an activity monitor (pedometer with accelerometer)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Arigo, Ph.D., Principal Investigator — Rowan University
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and analysis plan will be available via Open Science Framework (osf.io).
Supporting Information: Study Protocol, SAP
Time Frame: To be posted by 6/1 and accessible indefinitely.
Access Criteria: Public
URL: https://osf.io/

REFERENCES:
- [Derived] Arigo D, Baga K, Folk AL, Haggerty K. Physical activity partners for women with cardiovascular disease risk: Proof-of-concept trial with daily assessment. Health Psychol. 2025 Sep 29:10.1037/hea0001554. doi: 10.1037/hea0001554. Online ahead of print. PMID 41021523
- See also: Project website — https://drarigo.wordpress.com/womens-health-study-project-whade/